CLINICAL TRIAL: NCT01830413
Title: Stenting for Symtomatic Intracranial Artery Stenosis Registry in China
Brief Title: Stenting for Symptomatic Intracranial Artery Stenosis Registry in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Doc., Beijing Tiantan Hospital
Other Study IDs: stent-2013
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Systematic Intracranial Artery Stenosis
Keywords: stent, systematic Intracranial artery stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stenting: cerebral artery stenting for systematic Intracranial artery stenosis

SUMMARY:
Stenting for systematic Intracranial artery stenosis is challenged recently, especially for safety. This registry is aimed to explore the safety profile during peri-operation period in Stenting procedures for systematic Intracranial artery stenosis in Chinese population in real world.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year old
* medical failure patient with systematic Intracranial artery stenosis
* More than 3 weeks after most recent ischemic stroke
* Digital Subtraction Angiography(DSA) showed ≥70% stenosis in target intracranial artery
* Imaging test within 1 week showed bad collateral circulation in target vessel area
* Diseased vessel diameter≥2mm, length <15mm, distal vessel is normal

Exclusion Criteria:

* Diffused intracranial stenosis
* Acute stroke or TIA within 3 weeks
* Pure penetrating branch stenosis showed by cerebral imaging
* Non-atherosclerosis pathology for the stenosis
* Intracranial hemorrhage in target vessel area within 6 weeks; or potential cardiac thrombus source
* Intracranial tumor, arterial aneurysm or intracranial arteriovenous malformation

  •>50% stenosis in extracranial carotid artery or vertebral artery in operation side; Known contradiction to heparin, aspirin, clopidogrel, anesthesia or contrast; hemoglobin <10g/dl，platelet count <100000
* Modified Rankin score ≥3 related to target vessel;
* INR(International Normalized Ratio)>1.5(irreversible），persist hemorrhage risk; life expectancy < 1year
* Pregnant or beast-feeding
* Not suitable for endovascular stenting judged by Indication Judgement Committee

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with systematic Intracranial artery stenosis for stenting procedure
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety during peri-operation period | 30 days after operation
  Stroke in target cerebral vessel or death within 30 days after stenting procedure for systematic Intracranial artery stenosis

SECONDARY OUTCOMES:
Recurrent stroke in 30days to 1 year after stenting in target vessel area. | 30days to 1 year after stenting
  Recurrent stroke in 30days to 1 year after stenting in target vessel area.
Successful recanalization rate right after stenting | right after stenting
Stent restenosis rate | Within 1 year after stenting
Ischemic stroke outside target vessel area | 30 days - 1 year after stenting
Cerebral haemorrhage | 30 days - 1year after
Myocardial infarction | within 1 year
non-stroke haemorrhage | within 1year
Death in 30 days- 1 year after stenting | 30 days- 1 year after stenting
disabled stroke | within 1year
Any stroke or death | within 1 year
Serious adverse event | within 1year
National Institutes of Health Stroke Scale score(NIHSS score) | at 30 days and 1 year after stenting
Modified Rankin score(mRS) | at 30 days and 1 year after stenting
MoCA scale score | at 30 days and 1 year after stenting
Life quality scale score | at 1 year after stenting

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, M.D., Study Chair — Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beiing, Beijing Municipality, China